CLINICAL TRIAL: NCT00995930
Title: A Multi-center, Randomized , Double Blind, Placebo-controlled, Study of the Safety, Tolerability, and Effects on Arterial Structure and Function of ACZ885 in Patients With Clinically Evident Atherosclerosis and Either T2DM or IGT
Brief Title: Safety & Effectiveness on Vascular Structure and Function of ACZ885 in Atherosclerosis and Either T2DM or IGT Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CACZ885I2206; 2009-014618-80
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2015-03-06 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Diabetes Mellitus, Type 2; Atherosclerosis; Prediabetic State
Keywords: Atherosclerosis,; Type 2 Diabetes Mellitus, T2DM,; Cardiovascular Diseases, ACZ885, impaired glucose tolerance, IGT, Canakinumab
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Atherosclerosis; Prediabetic State; Cardiovascular Diseases; Glucose Intolerance | interventions — canakinumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): subcutaneous (SQ) monthly
  Interventions: Drug: Placebo
- ACZ885 (Experimental): 150 mg SQ monthly
  Interventions: Drug: ACZ885

INTERVENTIONS:
Drug: ACZ885 — ACZ885 150 mg was administered subcutaneously once a month for 12 months.
  Other Names: Canakinumab
  Arms: ACZ885
Drug: Placebo — Matching placebo to ACZ885 was administered subcutaneously once a month for 12 months.
  Arms: Placebo

SUMMARY:
This study will evaluate the effect of ACZ885 on vascular function in patients with documented atherosclerotic disease and T2DM or IGT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known atherosclerotic disease and documented diagnosis of T2DM for ≤ 14 years OR IGT
* HbA1c between 6.0% and 10.0%
* On stable statin therapy or statin intolerant
* Patients who are eligible and able to participate in the study

Exclusion Criteria:

* Contraindications to MRI
* NYHA class IV Heart Failure
* NYHA class I - III heart failure with acute exacerbation in 3 months prior to screening
* Patients with type 1 diabetes
* Acute infections
* HsCRP > 30 mg/dL
* Aortic aneurysm ≥5cm

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2009-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (9):
- United States (2):
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Cincinnati, Ohio
- Novartis Investigative Site, Montreal, Quebec, Canada
- Germany (3):
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Neuss
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Jerusalem, Israel
- United Kingdom (2):
  - Novartis Investigative Site, Oxford, UK
  - Novartis Investigative Site, London

REFERENCES:
- [Derived] Choudhury RP, Birks JS, Mani V, Biasiolli L, Robson MD, L'Allier PL, Gingras MA, Alie N, McLaughlin MA, Basson CT, Schecter AD, Svensson EC, Zhang Y, Yates D, Tardif JC, Fayad ZA. Arterial Effects of Canakinumab in Patients With Atherosclerosis and Type 2 Diabetes or Glucose Intolerance. J Am Coll Cardiol. 2016 Oct 18;68(16):1769-1780. doi: 10.1016/j.jacc.2016.07.768. PMID 27737744

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were randomized in a 1:1 ratio to each treatment arm.
Groups:
- Placebo: SQ monthly
Period: Overall Study
Arm/Group | Placebo | ACZ885
Started | 94 | 95
Safety Analysis Set | 94 | 95
Pharmacokinetic (PK) Analysis Set | 0 | 95
Pharmacodynamic (PD) Analysis Set | 92 | 92
Imaging Analysis Set | 92 | 92
Completed | 73 | 67
Not Completed | 21 | 28
Not completed — Protocol deviation | 2 | 5
Not completed — Death | 0 | 1
Not completed — Administrative problems | 4 | 2
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Adverse Event | 11 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ACZ885 | Total
Number analyzed (Participants) | 94 | 95 | 189
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.9 (6.92) | 61.7 (7.85) | 61.8 (7.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 80 | 82 | 162

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events, Serious Adverse Events and Death
Description: Participants were monitored for adverse events, serious adverse events and death throughout the study.
Time Frame: 12 months
Population: Safety analysis set: The safety analysis set included all randomized participants who received at least one dose of study drug.
Measure: Number; unit: Number of participants
Arm/Group | Placebo | ACZ885
Number analyzed (Participants) | 94 | 95
Number of participants
  Adverse events (serious and non-serious) | 80 | 77
  Serious adverse events | 14 | 25
  Deaths | 0 | 1

2. Primary Outcome: Change From Baseline in Aortic Distensibility
Description: Two axial, ECG-gated, steady state free precession (SSFP) 'cine' images were acquired during breath-hold to determine aortic distensibility. The first image was obtained at the level of the right pulmonary artery through the ascending and proximal descending aorta and the second through the distal aorta below the diaphragm. Imaging of the aorta also enabled evaluation of the plaque burden and additional vascular function measures.
Time Frame: baseline, 3 months, 12 months
Population: Only participants from the imaging analysis set, who had evaluable data at both baseline and the given post-baseline time point, were included in the analysis for that post baseline time point. The imaging analysis set included randomized participants who received at least one dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: mmHg^-1
Arm/Group | Placebo | ACZ885
Number analyzed (Participants) | 92 | 92
mmHg^-1
  3 months, proximal ascending region (n=61,63) | -0.0001 (0.0001) | 0.0001 (0.0001)
  12 months, proximal ascending region (n=56,55) | -0.0001 (0.0001) | -0.0001 (0.0001)

3. Primary Outcome: Change From Baseline in Plaque Burden (Aortic Vessel Wall Area and Carotid Vessel Wall Area)
Description: For assessment of atherosclerotic plaque burden of the aorta, vessel wall images of the aorta were acquired with an ECG gated double-inversion recovery (black blood) fast spin echo sequence applied breath-holding. Using an oblique sagittal image of the aorta as a pilot, serial axial images were acquired to cover a section of the descending thoracic aorta. The midpoint of the right pulmonary artery in cross section was used as the anatomical reference for the first slice in baseline and follow-up scans. For assessment of the atherosclerotic plaque burden in the carotids, vessel wall images were acquired with an axial ECG gated PD (proton density) weighted black blood sequence. The carotid bifurcation was used as the anatomical reference for all three imaging time points (baseline, 12 weeks, 48 weeks) with axial slice planes acquired below the bifurcation region. The mean values reported here for the carotid are reported for the proximal common carotid region.
Time Frame: baseline, 3 months, 12 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: mm^2
Arm/Group | Placebo | ACZ885
Number analyzed (Participants) | 92 | 92
mm^2
  aortic, proximal ascending, 3 months (n=69,62) | 14.80 (6.86) | -0.51 (6.62)
  aortic, proximal ascending, 12 months (n=61,53) | 30.58 (10.46) | 8.71 (10.49)
  carotid, mean (right and left), 3 months (n=66,59) | 1.41 (1.10) | -0.29 (1.12)
  carotid, mean (right and left), 12 mos. (n=55,48) | 3.50 (1.51) | 0.73 (1.48)

4. Secondary Outcome: Change From Baseline in Pulse Wave Velocity and Pulse Wave Velocity Error
Description: Utilizing the SphygmoCor Device, ECG leads placed at the carotid and femoral arteries provided the measure of the pulse wave at that particular arterial location. The distance between the two vascular beds divided by the pulse wave time shift provided a measure of the pulse wave velocity.
Time Frame: baseline, 3 months, 12 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ms^-1
Arm/Group | Placebo | ACZ885
Number analyzed (Participants) | 92 | 92
ms^-1
  pulse wave velocity, 3 months(n=45,38) | -0.39 (0.39) | -0.03 (0.39)
  pulse wave velocity, 12 months(n=35,31) | -0.36 (0.35) | -0.26 (0.35)
  pulse wave velocity error, 3 months (n=45,38) | -0.01 (0.05) | -0.03 (0.05)
  pulse wave velocity error, 12 months (n=35,31) | -0.01 (0.06) | 0.06 (0.06)

5. Secondary Outcome: Change From Baseline in Plaque Composition
Description: During the carotid MRI acquisition, in addition to the PD weighted ECG gated double inversion fast spin echo sequences T1 and T2 weighted sequences were acquired. In combination with the PD weighted images, the multi-contrast images were analyzed to determine regions of interest with contrast patterns consistent with the presence of necrotic lipid core, calcification and fibrous tissue in participants who had complex carotid plaque present in the bifurcation region.
Time Frame: baseline, 3 months, 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Placebo | ACZ885
Number analyzed (Participants) | 5 | 3
mm^2
  calcium composition, left carotid, 3 months | 0.002 (0.0045) | 0.003 (0.0058)
  calcium composition, left carotid, 12 months | 0.002 (0.0045) | 0.003 (0.0058)
  hemorrhage area, left carotid, 3 months | 0.006 (0.0114) | -0.000 (0.0200)
  hemorrhage area, left carotid, 12 months | 0.018 (0.0205) | 0.007 (0.0115)
  lipid composition, left carotid, 3 months | 0.000 (0.0000) | 0.003 (0.0115)
  lipid composition, left carotid, 12 months | -0.000 (0.0122) | 0.007 (0.0058)
  calcium composition,right carotid, 3 mos.(n=4,3) | -0.005 (0.0058) | -0.003 (0.0058)
  calcium composition,right carotid, 12 mos.(n=4,3) | 0.000 (0.0082) | 0.000 (0.0000)
  hemorrhage area,right carotid, 3 months (n=4,3) | 0.003 (0.0096) | -0.000 (0.0100)
  hemorrhage area, right carotid, 12 months (n=4,3) | 0.008 (0.0330) | 0.003 (0.0208)
  lipid composition, right carotid, 3 months (n=4,3) | -0.005 (0.0058) | 0.003 (0.0058)
  lipid composition, right carotid, 12 mos.(n=4,3) | 0.008 (0.0171) | 0.017 (0.0115)

6. Secondary Outcome: Change From Baseline in Aortic Strain
Description: Arterial strain was computed directly from the cine SSFP images and the change in lumen diameters over the cardiac cycle. The value was independent of pulse pressure and is unitless ratio derived from the maximum to minimum lumen diameters diastole and systole, respectively..
Time Frame: baseline, 3 months, 12 months
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | Placebo | ACZ885
Number analyzed (Participants) | 92 | 92
ratio
  proximal ascending, 3 months(n=67,64) | -0.005 (0.005) | 0.002 (0.005)
  proximal ascending, 12 months(n=59,59) | 0.001 (0.005) | -0.002 (0.005)

7. Secondary Outcome: Change From Baseline in High Sensitivity C-reactive Protein (hsCRP)
Description: Blood samples were collected to analyze hsCRP.
Time Frame: baseline, 3 months, 12 months
Population: Only participants from the PD analysis set, who had evaluable data at both baseline and the given post-baseline time point, were included in the analysis for that post baseline time point. The PD analysis set included randomized participants who received at least one dose of study medication.
Measure: Geometric Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Placebo | ACZ885
Number analyzed (Participants) | 92 | 92
mg/L
  3 months (n=82,79) | 0.93 [0.76 to 1.14] | 0.48 [0.39 to 0.58]
  12 months (n=73,68) | 1.04 [0.83 to 1.31] | 0.51 [0.41 to 0.64]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: Blood samples were collected to analyze fasting plasma glucose.
Time Frame: baseline, 3 months, 12 months
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | ACZ885
Number analyzed (Participants) | 92 | 92
mmol/L
  3 months (n=79,75) | 0.95 [0.89 to 1.01] | 1.00 [0.94 to 1.06]
  12 months (n=71,62) | 0.95 [0.87 to 1.02] | 0.99 [0.92 to 1.07]

9. Secondary Outcome: Change From Baseline in Hemoglobin A1c (HbA1c)
Description: Blood samples were collected to analyze HbA1c.
Time Frame: baseline, 3 months, 12 months
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: percentage
Arm/Group | Placebo | ACZ885
Number analyzed (Participants) | 92 | 92
percentage
  3 months (n=81,77) | 1.00 [0.97 to 1.02] | 0.99 [0.97 to 1.02]
  12 months (n=72,65) | 1.00 [0.96 to 1.04] | 0.96 [0.96 to 1.03]

10. Secondary Outcome: Change From Baseline in 2 Hour Glucose Post Oral Glucose Tolerance Test (OGTT)
Description: Blood samples were collected to analyze the 2 hour glucose post OGTT.
Time Frame: baseline, 3 months, 12 months
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo | ACZ885
Number analyzed (Participants) | 92 | 92
mmol/L
  3 months (n=79,74) | 0.92 [0.85 to 0.99] | 0.98 [0.90 to 1.05]
  12 months (n=71,62) | 0.93 [0.84 to 1.01] | 0.95 [0.88 to 1.04]

11. Secondary Outcome: Change From Baseline in Beta Cell Function (HOMA-B)
Description: Blood samples were collected to analyze beta cell function. Beta cell function was calculated by the Homeostasis Model Assessments (of beta cell function (HOMA-B) as follows: HOMA-B: The product of 20 and basal insulin (µU/mL) levels divided by the value of basal glucose (mmol/L) concentrations minus 3.5 [i.e., HOMA-B = 20*basal insulin/(basal glucose-3.5)].
Time Frame: baseline, 3 months, 12 months
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: percentage of beta cell function
Arm/Group | Placebo | ACZ885
Number analyzed (Participants) | 92 | 92
percentage of beta cell function
  HOMA-B, 3 months (n=77,70) | 1.11 [0.91 to 1.35] | 0.99 [0.82 to 1.20]
  HOMA-B, 12 months (n=71,60) | 1.03 [0.84 to 1.26] | 0.91 [0.75 to 1.10]

12. Secondary Outcome: Change From Baseline Insulin Resistance (HOMA-IR)
Description: Blood samples were collected to analyze insulin resistance. Insulin resistance was calculated by the Homeostasis Model Assessments of insulin resistance (HOMA-IR)) as follows: HOMA-IR: The product of basal glucose (mmol/L) and insulin (µU/mL) levels divided by 22.5 [i.e., HOMA-IR = basal glucose*basal insulin/22.5].
Time Frame: baseline, 3 months, 12 months
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: IR score
Arm/Group | Placebo | ACZ885
Number analyzed (Participants) | 92 | 92
IR score
  HOMA-R, 3 months (n=77,70) | 1.00 [0.85 to 1.18] | 1.09 [0.93 to 1.28]
  HOMA-R, 12 months (n=71,60) | 0.93 [0.77 to 1.13] | 0.97 [0.80 to 1.16]

13. Secondary Outcome: Pharmacokinetics: ACZ885 Serum Concentrations
Description: Blood samples were collected to analyze the ACZ885 serum concentrations.
Time Frame: pre-dose, 0.167 day post dose 1, 7 days post dose 1, 14 days post dose 1, every 30 days post each dose from doses 1 through 12, 60 days post dose 12, 90 days post dose 12
Population: Only participants from the PK analysis set, who had evaluable data at each time point, were included in the analysis for that time point. The PK analysis set included randomized participants from the ACZ885 arm who received at least one dose of study medication.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | ACZ885
Number analyzed (Participants) | 95
ng/mL
  pre-dose (n=91) | 0 (0)
  0.167 day post dose 1 (n=94) | 480 (648)
  7 days post dose 1 (n=95) | 10107 (4369)
  14 days post dose 1 (n=93) | 9138 (3527)
  30 days post dose 1 (n=90) | 5936 (2281)
  30 days post dose 2 (n=86) | 8136 (3299)
  30 days post dose 3 (n=81) | 9278 (3795)
  30 days post dose 4 (n=78) | 10183 (4552)
  30 days post dose 5 (n=78) | 10164 (4209)
  30 days post dose 6 (n=77) | 10254 (3916)
  30 days post dose 7 (n=76) | 10368 (4840)
  30 days post dose 8 (n=71) | 9745 (4436)
  30 days post dose 9 (n=69) | 10407 (3967)
  30 days post dose 10 (n=71) | 10635 (4697)
  30 days post dose 11 (n=70) | 10612 (4434)
  30 days post dose 12 (n=66) | 10887 (4785)
  60 days post dose 12 (n=66) | 4575 (2362)
  90 days post dose 12 (n=88) | 3241 (2883)

ADVERSE EVENTS:
Groups:
- ACZ885 150mg: ACZ885 150mg
Arm/Group | ACZ885 150mg | Placebo
Serious Adverse Events (participants affected / at risk) | 25/95 | 14/94
Other Adverse Events (participants affected / at risk) | 46/95 | 65/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 150mg (N=95) | Placebo (N=94)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina pectoris (Cardiac disorders) | 2 | 2
Angina unstable (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Epiglottitis (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty tophus (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACZ885 150mg (N=95) | Placebo (N=94)
Diarrhoea (Gastrointestinal disorders) | 5 | 6
Nausea (Gastrointestinal disorders) | 4 | 7
Vomiting (Gastrointestinal disorders) | 0 | 5
Asthenia (General disorders) | 2 | 5
Fatigue (General disorders) | 2 | 8
Influenza like illness (General disorders) | 4 | 5
Non-cardiac chest pain (General disorders) | 3 | 8
Nasopharyngitis (Infections and infestations) | 12 | 18
Upper respiratory tract infection (Infections and infestations) | 9 | 10
Blood creatine phosphokinase increased (Investigations) | 5 | 3
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 7
Dizziness (Nervous system disorders) | 5 | 5
Headache (Nervous system disorders) | 4 | 5
Renal failure (Renal and urinary disorders) | 2 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 6
Hypertension (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.